CLINICAL TRIAL: NCT04069585
Title: A Randomized, Controlled, Double-blinded, Within-subject (Split-face), Multicenter, Prospective Clinical Study to Compare the Level of Pain Using the Dermal Filler RHA® Redensity Formulated With Two Different Anesthetics in the Treatment of Perioral Rhytids
Brief Title: RHA® Redensity With New Anesthetic Agent - Perioral Rhytids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teoxane SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TEO-RHA-1801
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Results first posted 2021-06-16 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-05

CONDITIONS: Aging; Pain
Keywords: Hyaluronic Acid; Perioral rhytids; Anesthetic; Lidocaine
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Split-face design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- RHA® Redensity with new anesthetic agent (Experimental): Split-face injection of RHA® Redensity with new anesthetic agent in the perioral rhytids on one side of the mouth and RHA® Redensity with lidocaine in the perioral rhytids in the other side of the mouth.
  Up to 3 mL injected per side.
  Interventions: Device: RHA® Redensity with new anesthetic agent
- RHA® Redensity with lidocaine (Experimental): Split-face injection of RHA® Redensity with lidocaine in the perioral rhytids on one side of the mouth and RHA® Redensity with new anesthetic agent in the perioral rhytids in the other side of the mouth.
  Up to 3 mL injected per side.
  Interventions: Device: RHA® Redensity with lidocaine

INTERVENTIONS:
Device: RHA® Redensity with new anesthetic agent — A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus zooepidemicus, formulated to a concentration of 15 mg/g and 0.3% w/w of new anesthetic agent in a physiologic buffer.
  Arms: RHA® Redensity with new anesthetic agent
Device: RHA® Redensity with lidocaine — A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus zooepidemicus, formulated to a concentration of 15 mg/g and 0.3% w/w lidocaine in a physiologic buffer.
  Arms: RHA® Redensity with lidocaine

SUMMARY:
This is a randomized, controlled, double-blinded, within-subject (split-face), multicenter, prospective study to investigate whether RHA® Redensity with new anesthetic agent is non-inferior to RHA® Redensity with lidocaine in terms of injection site pain felt by the subject during injection.

At screening, the Treating Investigator (TI) evaluated subjects' perioral rhytid severity (using the Perioral Rhytid Severity Rating Scale; PR-SRS) to confirm eligibility and to establish a pre-treatment score for assessing aesthetic improvement.

At Visit 1, RHA® Redensity with new anesthetic agent was administered in a random sequence (first or second injection) and side of the mouth (left or right) and RHA® Redensity with lidocaine was administered to the other side. Study subjects and the TI injecting study devices were blinded.

Immediately after injection of an upper perioral quadrant, subjects rated the injection site pain experienced during injection using a 100 mm Visual Analog Scale (VAS). Injection site pain in each side of the mouth was also assessed at 15, 30, 45 and 60 minutes after injection of the upper quadrant.

Safety evaluation consisted of AE assessments, a 30-day CTR (Common Treatment Response) diary and a follow-up call performed by the study site at 72 hours after injection.

Subjects attended Visit 2 (30 days post-injection) where efficacy and safety assessments were conducted.

Subjects who presented with an unresolved clinically significant device related AE at Visit 2 received a optional follow-up phone call no later than 30 days after Visit 2.

If the clinically significant AE remained unresolved, the Investigator requested that the subject attended the optional in-clinic follow-up visit (i.e., Visit 3) within 5 working days. Follow-up of the clinically significant AE continued until the AE was resolved or the TI determines that additional follow-up was not necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient, male or female of any race, 22 years of age or older. Female subjects of childbearing potential must have a negative UPT at Visit 1 and practice a reliable method of contraception throughout the study.
2. Moderate to severe bilateral perioral rhytids (grade 2 or 3 on PR-SRS).
3. Perioral rhytids of the same PR-SRS grade on the left and right sides of the mouth.
4. Able to follow study instructions and complete all required visits.
5. Sign the IRB-approved ICF, Photographic Release Form, the Authorization for Use and release of Health and Research Study Information (HIPAA) form, and if applicable the California Experimental Research Subject's Bill of Rights prior to any study-related procedures being performed.

Exclusion Criteria:

1. Female subjects who are pregnant, breast-feeding, or of childbearing potential and not practicing reliable birth control.
2. Known hypersensitivity or previous allergic reaction to any component of the study devices.
3. Known sensitivity to local anesthetics of the amide type, history of multiple severe allergies, or history of anaphylactic shock.
4. Clinically significant active skin disease or infection in the perioral area within 6 months prior to study entry (TI discretion).
5. History of active chronic debilitating systemic disease that, in the opinion of the investigator, would make the subject a poor candidate in the study.
6. Malignancy (excluding non-melanoma skin cancer) within the past 5 years.
7. History or presence of condition or feature that may confound the interpretation of the results in the perioral region, for example, tattoo, significant facial hair, acne scaring, prior surgery in the area, potential for active disease or infection flare up such as herpes simplex.
8. History of skin cancer in the treatment area.
9. Elective, clinically significant facial procedures that may confound the interpretation of the results in the perioral region (TI discretion), prior to study enrollment.
10. Clinically active disease or infection in the perioral area or mouth (e.g., dental abscess).

12. Exposure to any other investigational drug/device within 90 days of entering the study.

13. Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - California, Beverly Hills, California
  - Florida, Coral Gables, Florida
  - Chicago, Chicago, Illinois

REFERENCES:
- [Derived] Kaufman-Janette J, Joseph JH, Dayan SH, Smith S, Eaton L, Maffert P. Patient Comfort, Safety, and Effectiveness of Resilient Hyaluronic Acid Fillers Formulated With Different Local Anesthetics. Dermatol Surg. 2022 Oct 1;48(10):1065-1070. doi: 10.1097/DSS.0000000000003541. Epub 2022 Jul 13. PMID 36129233

RESULTS

PARTICIPANT FLOW:
Groups:
- Bilateral Treatment RHA® Redensity With New Anesthetic Agent Vs RHA® Redensity With Lidocaine: Split-face injection of RHA® Redensity With New Anesthetic Agent in the perioral rhytids on one side of the mouth and RHA® Redensity with lidocaine in the perioral rhytids on the other side of the mouth.
  RHA® Redensity With New Anesthetic Agent was administered in a random sequence (first or second injection) on one side of the mouth and RHA® Redensity with lidocaine was administered in the other side.
Period: Overall Study
Arm/Group | Bilateral Treatment RHA® Redensity With New Anesthetic Agent Vs RHA® Redensity With Lidocaine
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Bilateral Treatment With RHA® Redensity With New Anesthetic Agent Vs RHA® Redensity With Lidocaine: Split-face injection of RHA® Redensity With New Anesthetic Agent in the perioral rhytids on one side of the mouth and RHA® Redensity with lidocaine in the perioral rhytids on the opposite side of the mouth.
Arm/Group | Bilateral Treatment With RHA® Redensity With New Anesthetic Agent Vs RHA® Redensity With Lidocaine
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick scale is a numerical classification schema for human skin color.
  Type I - always burns, never tans (pale white; blond or red hair; blue eyes; freckles).
  Type II - usually burns, tans minimally (white; fair; blond or red hair; blue, green, or hazel eyes) Type III - sometimes mild burn, tans uniformly (cream white; fair with any hair or eye color) Type IV - burns minimally, always tans well (moderate brown) Type V - very rarely burns, tans very easily (dark brown) Type VI - Never burns, never tans (deeply pigmented dark brown to darkest brown)
  Participants
    Types I to III as assessed by TI at screening | 23
    Types IV to VI as assessed by TI at screening | 7

OUTCOME MEASURES:

1. Primary Outcome: Non-inferiority of RHA® Redensity With New Anesthetic Agent Versus RHA® Redensity With Lidocaine in Terms of Reducing Pain During Device Injection Into the Upper Perioral Rhytids.
Description: Injection pain during injection was measured on the 100 mm Visual Analog Scale (VAS), as assessed by subjects immediately after injection of each upper perioral quadrant.
  VAS is a 100 mm Visual Analog Scale with 0 meaning no pain and 100 meaning intolerable pain
Time Frame: Visit 1 - During Injection
Population: There were 30 participants enrolled and treated, the participants received bilateral, split-face treatment into the upper perioral rhytids.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- RHA® Redensity With New Anesthetic Agent: RHA® Redensity with new anesthetic agent A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus zooepidemicus, formulated to a concentration of 15 mg/g and 0.3% w/w of a new anesthetic agent in a physiologic buffer.
Arm/Group | RHA® Redensity With Lidocaine | RHA® Redensity With New Anesthetic Agent
Number analyzed (Participants) | 30 | 30
mm | 22.4 (23.21) | 25.0 (25.63)
Statistical Analysis 1: Comparison: RHA® Redensity With Lidocaine vs RHA® Redensity With New Anesthetic Agent; Test type: Non-Inferiority — To achieve non-inferiority, the observed p-value must be <= 0.5 taking into account of the non-inferiority margin (i.e., 10mm difference in Pain VAS between the two treatment groups); p < 0.0002, t-test, 1 sided — One-sided paired t-test

2. Secondary Outcome: Difference Between RHA® Redensity With New Anesthetic Agent Versus RHA® Redensity With Lidocaine in Term of Reducing Pain at 15, 30, 45 and 60 Minutes Post-injection in Each Side of the Mouth.
Description: Injection pain was measured on the 100 mm Visual Analog Scale (VAS), as assessed by subjects in each side of the mouth.
  VAS is a 100 mm Visual Analog Scale with 0 meaning no pain and 100 meaning intolerable pain
Time Frame: Visit 1 - 15, 30, 45 and 60 minutes post-injection
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | RHA® Redensity With Lidocaine | RHA® Redensity With New Anesthetic Agent
Number analyzed (Participants) | 30 | 30
mm
  15 Min | 6.3 (12.29) | 6.8 (13.72)
  30 Min | 1.0 (4.03) | 1.0 (4.19)
  45 Min | 0.3 (1.83) | 0.4 (2.37)
  60 Min | 0.0 (0.00) | 0.0 (0.00)

3. Secondary Outcome: Change From Baseline of PR-SRS Score for RHA® Redensity With New Anesthetic Agent Vs RHA® Redensity With Lidocaine for the Correction of Perioral Rhytids as Assessed by the Treating Investigator (TI)
Description: PR-SRS (Perioral Rhytids Severity Rating Scale) is a validated 4-grade scale with 0 being "Absent" and 3 being "Severe"
Time Frame: Visit 1 (Baseline, pre-injection) - Visit 1 (post-injection), Visit 2 (Day 30)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RHA® Redensity With Lidocaine | RHA® Redensity With New Anesthetic Agent
Number analyzed (Participants) | 30 | 30
units on a scale
  Visit 1 (Post-injection) | -1.5 (0.57) | -1.5 (0.63)
  Visit 2 (Day 30) | -1.4 (0.57) | -1.4 (0.56)

4. Secondary Outcome: Percentage of Responders Based on the Intra-individual Improvement of at Least One Grade on the Perioral Rhytids Severity Rating Scale (PR-SRS) Compared to Baseline, as Assessed by the TI
Description: A responder corresponds to a subject with an intra-individual improvement of at least one grade on the PR-SRS compared to Baseline
Time Frame: Visit 1 - Baseline (pre-injection), Visit 1 (post-injection), Visit 2 (Day 30)
Measure: Count of Participants; unit: Participants
Arm/Group | RHA® Redensity With Lidocaine | RHA® Redensity With New Anesthetic Agent
Number analyzed (Participants) | 30 | 30
Participants
  Visit 1 - post-injection: Responder | 29 | 28
  Visit 1 - post-injection: Not responder | 1 | 2
  Visit 2 - day 30: Responder | 29 | 29
  Visit 2 - day 30: Not responder | 1 | 1

5. Secondary Outcome: Subject's Perception of Treatment Effectiveness as Per the FACE-Q (Perioral Rhytids Domain) Questionnaire.
Description: The FACE-Q measures the experience and outcomes of aesthetic facial procedures from the patient's perspective.
  FACE-Q questionnaire is composed of 6 questions with a score linked to answers (1 being 'Not at all' and 4 being 'Extremely').
  The subject will be instructed as follows: ""These questions ask about how you look right now. For each question, circle only one answer. With the area around your lips in mind, in the past week, how much have you been bothered by:", and will provide response.
  To calculate the FACE-Q, outcomes from all 6 questions were pooled, data were transformed so that higher scores reflected a superior outcome, and adapted to a scale of 100 units (i.e. lowest score = 0, highest score = 100).
Time Frame: Visit 1 (Baseline) and Visit 2 (Day 30)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RHA® Redensity With Lidocaine | RHA® Redensity With New Anesthetic Agent
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline Face-Q Score | 13.0 (19.07) | 12.5 (18.99)
  Day 30 Face-Q Score | 73.9 (28.84) | 77.2 (25.78)
  Face-Q Change from Baseline to Day 30 | 60.9 (36.10) | 64.7 (31.93)

6. Secondary Outcome: Number of Subjects Scored Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) by the Treating Investigator (TI)
Description: Global Aesthetic Improvement (GAI) is a subjective 5-grade scale comprised of "much improved, improved, no change, worse, and much worse".
  GAI will bewas assessed using the baseline photograph. Each side of the mouth were assessed independently.
Time Frame: Visit 1 (post-injection) and Visit 2 (Day 30)
Measure: Count of Participants; unit: Participants
Arm/Group | RHA® Redensity With Lidocaine | RHA® Redensity With New Anesthetic Agent
Number analyzed (Participants) | 30 | 30
Participants
  Visit 1 (post-injection) | 30 | 30
  Visit 2 (Day30) | 30 | 30

7. Secondary Outcome: Number of Global Aesthetic Improvement (GAI) Responders (i.e., Scoring Either "Much Improved" or "Improved") on GAI Scale According to Subject's Self-assessment
Description: Global Aesthetic Improvement (GAI) is a subjective 5-grade scale comprised of "much improved, improved, no change, worse, and much worse".
  GAI was assessed using the baseline photograph. Subjects were instructed as follows: "Use a mirror to compare your face to the photograph provided to you and rate the degree of aesthetic improvement by using the following scale".
  Each side of the face was assessed independently.
Time Frame: Visit 1 (post-injection) and Visit 2 (Day 30)
Measure: Count of Participants; unit: Participants
Arm/Group | RHA® Redensity With Lidocaine | RHA® Redensity With New Anesthetic Agent
Number analyzed (Participants) | 30 | 30
Participants
  Visit 1 (post-injection) | 30 | 30
  Visit 2 (Day 30) | 30 | 30

8. Secondary Outcome: Number of Both "Satisfied" or "Very Satisfied" Subjects With Study Treatment Using the Subject's Satisfaction Scale
Description: The Subject Satisfaction Scale is a subjective, balanced, 5-point scale assessing subject satisfaction with study treatment. Possible scores range from with 1 (very satisfied) to 5 (very dissatisfied).
  Proportion of subjects who were Satisfied (i.e., 1-Very Satisfied + 2-Satisfied) was compared to the proportion of subjects who were Not Satisfied (i.e., 3-Neither Satisfied nor dissatisfied + 4-Dissatisfied + 5-Very Dissatisfied)
Time Frame: Visit 1 (post-injection) and Visit 2 (Day 30)
Measure: Count of Participants; unit: Participants
Arm/Group | RHA® Redensity With Lidocaine | RHA® Redensity With New Anesthetic Agent
Number analyzed (Participants) | 30 | 30
Participants
  Visit 1 (post-injection): Satisfied (i.e., 1-Very Satisfied + 2-Satisfied) | 29 | 29
  Visit 1 (post-injection): Not Satisfied (i.e., 3-Neither Satisfied nor dissatisfied + 4-Dissatisfied + 5-Very Dissatisfied) | 1 | 1
  Visit 2 (Day 30): Satisfied (i.e., 1-Very Satisfied + 2-Satisfied) | 29 | 29
  Visit 2 (Day 30): Not Satisfied (i.e., 3-Neither Satisfied nor dissatisfied + 4-Dissatisfied + 5-Very Dissatisfied) | 1 | 1

9. Secondary Outcome: Number of Subjects With Post Injection Treatment Responses (From Common Treatment Responses (CTR) Diary) for Safety Evaluation of RHA® Redensity With New Anesthetic Agent Versus RHA® Redensity With Lidocaine
Description: The subjects will receive a diary booklet and instructions for recording his/her observations of the Common Treatment Responses to the study treatments within 30 days following the treatment. The diary will be discussed during follow-up phone-call and visit. Subjects were instructed to complete the diary at approximately the same time each day (i.e., am or pm).
  The subject diary captured the following Common Treatment Responses (CTR) that occur following the injection of a dermal filler; specifically, redness, pain, tenderness, firmness, swelling, lumps/bumps, bruising, itching, discoloration, and "other".
  The 30-day patient CTR diary included a detailed glossary describing all signs/symptoms listed in the diary; an option was provided to report "other" reactions if the subject experienced a sign/symptom that was not listed.
Time Frame: During 30 days after injection
Measure: Count of Participants; unit: Participants
Arm/Group | RHA® Redensity With Lidocaine | RHA® Redensity With New Anesthetic Agent
Number analyzed (Participants) | 30 | 30
Participants
  Bruising | 16 | 12
  Discoloration | 10 | 10
  Firmness | 19 | 14
  Itching | 2 | 4
  Lumps/Bumps | 17 | 15
  Pain | 4 | 3
  Redness | 15 | 16
  Swelling | 19 | 21
  Tenderness | 12 | 13
  Needle track marks | 1 | 1
  Injection Site Soreness | 1 | 1

ADVERSE EVENTS:
Time Frame: 1 month (33 days, overall study duration)
Arm/Group | RHA® Redensity With New Anesthetic Agent | RHA® Redensity With Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/30
Other Adverse Events (participants affected / at risk) | 6/30 | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RHA® Redensity With New Anesthetic Agent (N=30) | RHA® Redensity With Lidocaine (N=30)
Osteomyelitis (toe on left foot) (Infections and infestations) | 1 (1) | 1 (1) — Osteomyelitis (toe on left foot) diagnosed in one patient, which underwent amputation of the affected toe - The event was unrelated to the study devices. SAE outcome was deemed to be resolved within 6 days.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RHA® Redensity With New Anesthetic Agent (N=30) | RHA® Redensity With Lidocaine (N=30)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 1 (1)
Injection site induration (General disorders) | 2 (4) | 2 (2)
Injection site mass (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (2) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Needle track marks (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT04069585/Prot_002.pdf
  • Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT04069585/SAP_003.pdf